CLINICAL TRIAL: NCT06124781
Title: The Value of Molecular Signatures in the Diagnosis of Allergic Contact Dermatitis.
Brief Title: Molecular Diagnosis of Allergic Contact Dermatitis (SMECA).
Acronym: SMECA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00231-40
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Eczema; Allergic Contact Eczema Nos
MeSH Terms: conditions — Eczema | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with patch test reactions (Experimental): Patient with at least one positive/doubtful patch test reaction for nickel, limonene hydroperoxide and/or linalool hydroperoxide
  Interventions: Procedure: Blood sample; Procedure: Skin biopsies; Procedure: ROAT test

INTERVENTIONS:
Procedure: Blood sample — A blood sample (48 ml) will be collected from each patient before performing the ROAT tests. This sample will be used to perform in vitro lymphocyte proliferation test, and cytokine measurements.
Procedure: Skin biopsies — 2 skin biopsies will be performed at the inclusion: one from positive/doubtful patch test reaction and one from control patch test. In case of positive ROAT test, 2 additional biopsies will be collected: one from positive ROAT test reaction and one from control area. Molecular analysis will be performed.
Procedure: ROAT test — ROAT test (repeated open application test) is a use test used to establish the clinical relevance of patch tests. Patients will be exposed to 3 solutions of increasing concentration containing the culprit allergen (nickel, limonene hydroperoxide or linalool hydroperoxide), as well as a solution containing the vehicle alone (control solution), 2 times a day for up to 21 days, in the absence of a reaction.

SUMMARY:
Allergic contact dermatitis (ACD) is a common inflammatory skin disease, which represents a major public health issue in industrialized countries. ACD is induced by repeated contact of individuals with environmental chemicals and is characterized by a delayed type IV hypersensitivity response with skin inflammation mediated by allergen-specific T cells in sensitized individuals.

The current diagnosis is based on clinical examination, assessment of environmental exposures and patch testing. Although the robustness of patch tests has long been established, this method can sometimes give inconclusive results, leading to problems in disease management.

Preliminary results indicate that the molecular analysis of Patch-Tests (PT) reactions could allow a more reliable diagnosis. Importantly, this gene profiling approach may help to identify patients with false positive PT reactions, i.e. patients whose PT reactions did not show any "allergy signature".

However, it remains to be demonstrated that the presence or absence of allergy biomarkers in PT lesions are indeed predictive of ACD response in patients.

The main objective is to describe the correlation between these molecular signatures and the reactivity of individuals when they are exposed to allergenic compounds under conditions of use (using ROAT test).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age.
* Patient with at least one positive/doubtful patch test reaction for nickel, limonene hydroperoxide and/or linalool hydroperoxide
* Patient agreeing to undergo skin biopsies and blood sampling
* Patient agreeing to non-identifying pictures being taken of lesions
* Patient available to carry out skin tests and their interpretation
* Patient affiliated to or benefiting from a social security regime
* Patient having been informed and having signed a written, free and informed consent.

Exclusion Criteria:

* Patient with active dermatitis lesions on the forearm
* Patient with a history of allergic reaction to a local anesthetic product
* Patient with wound healing disorders (hypertrophic or keloids scars)
* Patient with hematological disorders
* Patient having topical treatments with corticosteroids or immunomodulators on the forearms during the 21 days prior to the start of the study
* Patient having had excessive exposure to ultraviolet during the 21 days prior to the start of the study.
* Patient on systemic corticosteroid therapy, immunosuppressants or biological therapy.
* Patient whose follow-up is impossible for reasons psychological or geographical.
* Patient taking part in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breast-feeding or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Expression levels of allergy biomarkers | 1 month
  Expressed as fold change (ratio between gene expression levels in lesional skin of patch test reaction and their expression levels in healthy skin = control patch test, of the same patient) in patients with positive or negative ROAT test (Gold standard)

CONTACTS AND LOCATIONS:
Locations (5):
- Clinique universitaire Saint Luc, Brussels, Belgium
- France (4):
  - CHU de Grenoble, La Tronche
  - CHU Lyon Sud, Pierre-Bénite
  - Hopital Privé de la Loire, Saint-Etienne
  - CHU de Saint Etienne, Saint-Priest-en-Jarez

REFERENCES:
- [Result] Nosbaum A, Vocanson M, Rozieres A, Hennino A, Nicolas JF. Allergic and irritant contact dermatitis. Eur J Dermatol. 2009 Jul-Aug;19(4):325-32. doi: 10.1684/ejd.2009.0686. PMID 19447733
- [Result] Vocanson M, Hennino A, Chavagnac C, Saint-Mezard P, Dubois B, Kaiserlian D, Nicolas JF. Contribution of CD4(+ )and CD8(+) T-cells in contact hypersensitivity and allergic contact dermatitis. Expert Rev Clin Immunol. 2005 May;1(1):75-86. doi: 10.1586/1744666X.1.1.75. PMID 20477656
- [Result] Vocanson M, Hennino A, Rozieres A, Poyet G, Nicolas JF. Effector and regulatory mechanisms in allergic contact dermatitis. Allergy. 2009 Dec;64(12):1699-714. doi: 10.1111/j.1398-9995.2009.02082.x. Epub 2009 Oct 12. PMID 19839974
- [Result] Lefevre MA, Nosbaum A, Rozieres A, Lenief V, Mosnier A, Cortial A, Prieux M, De Bernard S, Nourikyan J, Jouve PE, Buffat L, Hacard F, Ferrier-Lebouedec MC, Pralong P, Dzviga C, Herman A, Baeck M, Nicolas JF, Vocanson M. Unique molecular signatures typify skin inflammation induced by chemical allergens and irritants. Allergy. 2021 Dec;76(12):3697-3712. doi: 10.1111/all.14989. Epub 2021 Jul 14. PMID 34174113
- [Result] Ljungberg Silic L, Lefevre MA, Bergendorff O, De Bernard S, Nourikyan J, Buffat L, Nosbaum A, Bruze M, Nicolas JF, Svedman C, Vocanson M. Gene profiling reveals a contact allergy signature in most positive Amerchol L-101 patch test reactions. Contact Dermatitis. 2022 Jul;87(1):40-52. doi: 10.1111/cod.14077. Epub 2022 Mar 25. PMID 35184302